CLINICAL TRIAL: NCT04280055
Title: Prophylactic Effects of Psilocybin on Chronic Cluster Headache: an Open-label Clinical Trial and Neuroimaging Study
Brief Title: Prophylactic Effects of Psilocybin on Chronic Cluster Headache
Acronym: EPOCH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not possible to achieve the anticipated no. of patients due to Covid-19 pandemic
Sponsor: Gitte Moos Knudsen (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Chair, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-18040896
Record Dates: First submitted 2020-02-12; First posted 2020-02-21 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cluster Headache
Keywords: Cluster Headache; Psilocybin; Prophylactic; Treatment; Hallucinogens
MeSH Terms: conditions — Cluster Headache | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 0.14 mg/kg p.o. in three sessions spaced by one week

SUMMARY:
The purpose of this study is to investigate the prophylactic effects of psilocybin in chronic cluster headache. Subjects will receive a low dose of psilocybin during 3 sessions spaced by one week. Subjects will maintain a headache diary prior to, during, and after the administrations in order to document headache frequency, intensity and duration. Subjects will undergo a fMRI scanning before the first and after the last psilocybin session.

DETAILED DESCRIPTION:
Cluster headache (CH) is one of the most painful conditions known. CH affects 1 out 1000 and exists in two well-defined forms: episodic (ECH) and chronic (CCH). Ten to fifteen percent of patients have CCH and have less than three months of pain-free time during a year. Medical treatment for CH is divided into acute abortive treatment for the single attack and a prophylactic treatment. The most commonly used prophylactic, verapamil, decreases attack frequency but does not induce remission and very high doses are needed. Although most therapeutic options ameliorate CH, they may be problematic due to major side effects, unsatisfactory treatment response or availability. Thus, novel treatment options are needed. According to several studies, patients that self-medicate with low doses of the serotonin 2A receptor (5-HT2AR) agonist and psychedelic psilocybin report that this is effective as CH prophylaxis or even to induce remission. So far, no clinical trials to confirm this have been conducted, nor is there any objective measures of brain function in association with psilocybin intake in CH. There is, however, already some evidence from functional magnetic resonance (fMRI) imaging studies suggesting that CH patients have abnormal functional connectivity patterns involving the hypothalamus and distributed brain networks, but the implication of these abnormalities is unknown.

The investigators are conducting a prospective pilot study, evaluating prophylactic effects of psilocybin in CCH using an open-label study design. They're also going to investigate psilocybin's active metabolite psilocin and brain function (fMRI) to identify possible brain mechanisms underlying CCH and treatment response, including the correlation of treatment response with psilocin levels and estimated 5-HT2AR occupancy and the extent to which brain network changes are affected by psilocybin and correlated with treatment response.

Effects of psilocybin on headache frequency, duration and intensity will be assessed in a sample of 20 patients with CCH. Participants will fill out headache logs during the entire study period, in total 10 weeks. Before study inclusion, participants taking prophylactic medication will first go through a 2-week wash-out period to allow for elimination of the medicine. Inclusion is followed by a baseline observation period lasting four weeks, after which patients will first undergo a baseline rs fMRI scanning followed by the first dose of 0.14 mg/kg psilocybin p.o. Blood samples will be collected during the first psilocybin intervention to establish psilocin plasma concentrations, which will be used for estimating receptor occupancy. Participants will then undergo two additional psilocybin administrations spaced by one-week. The last psilocybin dose will be followed by 4 weeks of observation. One week after the last administration of psilocybin, participants will undergo a follow-up MRI scan. Participants will be contacted 3, 6 and 12 months after the last psilocybin dose to gain information about the duration of potential remission periods. All regular acute treatments are permitted during the study period and a systematic record hereof has to be noted in the headache diary. No other prophylactic medication is allowed during the trial and at least a two-week washout period before inclusion is required. Prophylactics are allowed again after the 4 weeks follow-up, with dose and type carefully recorded. Participants will fill out questionnaires during the observation period, in conjunction with psilocybin interventions and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* A diagnosis of chronic cluster headache according to IHCD-III.
* Ability to separate cluster headache attacks from other types of headache.
* A history of at least 4 attacks/week in the last 4 weeks before inclusion

Exclusion Criteria:

* A history of using a serotonergic hallucinogen for CH.
* Participation in any clinical trials within 30 days preceding study enrollment.
* Use of other prophylactic CH medication within the last two weeks.
* Current use of drugs suspected to interfere with treatment (e.g. antipsychotic medication) or to be hazardous in combination with psilocybin.
* Presence of other trigeminal autonomic cephalalgias.
* Known hypersensitivity/allergy to multiple drugs (including psilocybin).
* A history or presence of any medical and psychiatric condition that might render patient unsuitable for participation.
* Present or previous manic or psychotic disorder or critical psychiatric disorder.
* Current drug or alcohol abuse.
* MRI Contraindications.
* Pregnancy or breastfeeding
* Not using safe contraception (if fertile woman)
* Stroke (<1 year from inclusion)
* Myocardial infarction (<1 year from inclusion)
* Hypertension (> 140/90 mmHg at inclusion)
* Clinically significant arrhythmia (<1 year from inclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Week 6-10 (post drug observation) compared to week 0-4 (baseline observation)
  Change in headache frequency in number of attacks/week
Resting state FC fMRI analyses | Day 1 of first psilocybin session to 1 week after last psilocybin session (3 weeks)
  Resting state FC fMRI analyses, including hypothalamic FC, comparing baseline and rescan, comparison with healthy control sample, and evaluation of correlation between headache frequency changes and FC changes.

SECONDARY OUTCOMES:
Proportion of reduced frequency | Week 6-10 (post drug observation) compared to week 0-4 (baseline observation)
  Proportion of patients with a 50% reduction in headache frequency
Headache intensity | Week 6-10 (post drug observation) compared to week 0-4 (baseline observation)
  Change in average headache intensity of attacks (0-10 on Visual Analog Scale (VAS), where 0 is no pain and 10 is worst pain imaginable)
Need of acute therapy | Week 6-10 (post drug observation) compared to week 0-4 (baseline observation)
  Number of attacks requiring acute therapy
Sideeffects | Whole observation period (10 weeks)
  Proportion of patients experiencing serious side effects
Remission | Day 1 after first psilocybin session until 12 month follow up (1 year).
  Proportion of patients with remission lasting more than 1 month
Remission duration | Day 1 after first psilocybin session until 12 month follow up (1 year).
  Duration of induced remission (number of weeks)
SF-36 | Week 6-10 (post drug observation) compared to week 0-4 (baseline observation)
  Quality of life assessed by questionnaires: The Short Form (36) Health Survey. SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Preferred treatment | Whole observation period (10 weeks)
  Proportion of patients that prefers to continue with psilocybin if this was an option or want to return to usual prophylactics.
Mood | Pre-psilocybin (week 1 and 5) vs post-psilocybin (week six and eight).
  Changes in mood measured be the POMS questionaire.
Sleep quality | Pre-psilocybin (week 1 and 5) vs post-psilocybin (week six and eight).
  Sleep quality measured by the PSQI questionaire.
Depressive symptoms | Pre-psilocybin (week 1 and 5) vs post-psilocybin (week six and eight).
  Depressive symptoms measured by the MDI questionaire.
Stress | Pre-psilocybin (week 1 and 5) vs post-psilocybin (week six and eight).
  Perceived stress measured by the PSS questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Moos Knudsen, MD, DMSc, Study Chair — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for integrated Molecular Brain Imaging (CIMBI) data will be available for neuroscience research community contingent on approval by scientific board.

REFERENCES:
- See also: Online preprint of the outcome of the study. Positive! — https://www.medrxiv.org/content/10.1101/2022.07.10.22277414v1